CLINICAL TRIAL: NCT06710392
Title: Evaluate the Safety and Efficacy of Two Enzyme Cocktails in Healthy Adults With Subclinical Mild to Moderate Gastrointestinal Complaints
Brief Title: Efficacy of Two Enzyme Cocktails in Healthy Adults
Acronym: ElZyme
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: University of North Texas, Denton, TX (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CTB2022TN225D
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Digestive; Gastrointestinal Health
Keywords: enzyme; enzyme cocktail; healthy adults; nutraceutical

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Digestive Enzyme Cocktail A (Experimental): Arm receiving investigational product A
  Interventions: Dietary Supplement: Enzyme Cocktail A
- Digestive Enzyme Cocktail B (Experimental): Arm receiving investigational product B
  Interventions: Dietary Supplement: Enzyme Cocktail B
- Placebo A (Placebo Comparator): Arm receiving placebo A
  Interventions: Dietary Supplement: Placebo A
- Placebo B (Placebo Comparator): Arm receiving Placebo B
  Interventions: Dietary Supplement: Placebo B

INTERVENTIONS:
Dietary Supplement: Enzyme Cocktail A — Enzyme cocktail A in the form of a capsule with a daily dose of 275mg taken 3 times a day for 4 weeks.
  Arms: Digestive Enzyme Cocktail A
Dietary Supplement: Enzyme Cocktail B — Enzyme cocktail B in the form of a capsule with a daily dose of 50mg taken 3 times a day for 4 weeks.
  Arms: Digestive Enzyme Cocktail B
Dietary Supplement: Placebo A — Placebo A matching investigational product A given 3 times a day for 4 weeks.
  Arms: Placebo A
Dietary Supplement: Placebo B — Placebo B matching investigational product B given 3 times a day for 4 weeks.
  Arms: Placebo B

SUMMARY:
The goal of this study is to determine the safety and efficacy of two enzyme cocktails in healthy adults with mild to moderate gastrointestinal discomfort. The main question aims to answer whether a 4-week administration of an enzyme cocktail can improve how the participant feels about their gut health. This is done by completing a weekly questionnaire, and the results are compared between the 4 weeks the participants are on a placebo and the 4 weeks the participants are on the enzyme cocktail. Participants will also provide a stool sample at the start and end of each treatment. Stool samples will collected and stored in case further microbiome analysis is warranted.

ELIGIBILITY:
Exclusion Criteria:

* Presence of a serious congenital anomaly or chronic medical condition that would contraindicate participation, including history of major gastrointestinal surgery, chronic gastrointestinal illness, abnormal intestinal anatomy or significant abdominal disorder
* Having taken oral antibiotics in the previous 3-months or if they start antibiotics during the study
* Currently or having taken a prebiotic, probiotic, or digestive enzyme supplement in the previous 3-months
* Currently consuming 1 or more servings of fermented foods or yogurt on a daily basis
* Doctor diagnosed chronic disease (i.e. Diabetes, Cardiovascular, etc.)
* Doctor diagnosed immunodeficiency
* Current use of doctor prescribed immunosuppressive agents (corticosteroids, methotrexate, etc.)
* Pregnancy, 6 months postpartum period, or current breastfeeding
* Women of childbearing age planning pregnancy during the course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Gastrointestinal Symptoms Rating Scale - Irritable Bowel Syndrome (GSRS-IBS) | From baseline to the end of intervention 4 weeks later.
  Change in GSRS-IBS total score from baseline to end of intervention. Each question is rated on a 7 point Likert scale with higher scores representing more troublesome symptoms. Questionnaire collected weekly from baseline through study completion at the end of week 12.

SECONDARY OUTCOMES:
Change from baseline in Stool Consistency at end of intervention | Through study completion, an expected average of 70 days
  Difference in weekly self reported stool consistency, as measured by the Bristol Stool Form Scale (BSFS) on a daily basis. BSFS max score 7 - lower scores indicate constipation, higher scores indicate diarrhea.
Change from baseline in the Stool Frequency at end of intervention | Through study completion, an expected average of 70 days
  Change in weekly average stool frequency throughout the period between baseline and end of intervention.
Change in Microbiome (faecal samples) | Day 0 and Day 28; Day 42 and Day 70
  Change in stool microbiome between baseline and end of intervention for each of cross over runs (Change between day 0 and day 28, change between day 42 and 70)
Body Mass Index (BMI) | Day 0, Day 28, Day 42, and Day 70
  Participants whole-body weight [kg] and height [m] will be measured and BMI will be calculated as kg/m^2
Total Fat Mass | Day 0, Day 28, Day 42, and Day 70
  Participants total fat mass (kg) will be tested using a BIA scale.
Food Intake | Day 0
  Food intake is measured by the NHANES Food Frequency Questionnaire (NHANES-FFQ), which collects data to measure habitual food intake at baseline.
Positive and Negative Affect Schedule (PANAS-SF) | Day 0, Day 28, Day 42, and Day 70
  The PANAS-SF is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of North Texas, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No